CLINICAL TRIAL: NCT01796353
Title: A Randomized Clinical Trial of a Comprehensive Sexual Rehabilitation Programme Versus Usual Care in Male Patients With Impaired Sexual Function and Ischemic Heart Disease or Implantable Cardioverter Defibrillator
Brief Title: Effects of a Comprehensive Sexual Rehabilitation Programme in Heart Patients
Acronym: CopenHeartSF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Researcher, Ph.D, post.doc., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CopenHeart-SF
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Ischaemic Heart Disease; Cardiac Arrhythmia; Sexual Dysfunction
Keywords: heart disease; sexual dysfunction; exercise test; comprehensive rehabilitation; complex intervention
MeSH Terms: conditions — Coronary Artery Disease; Arrhythmias, Cardiac; Sexual Dysfunction, Physiological; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sexual rehabilitation (Experimental): exercise plus psycho-education
  Interventions: Other: sexual rehabilitation
- usual care (Active Comparator): usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: sexual rehabilitation — exercise plus psycho-education
  Arms: sexual rehabilitation
Other: Usual care — usual care
  Arms: usual care

SUMMARY:
The objective is to investigate the effect of a comprehensive sexual rehabilitation program, consisting of a psycho-educative component and a physical exercise component.

The primary hypothesis is that, a comprehensive sexual rehabilitation program improves sexual function.

DETAILED DESCRIPTION:
Sexual function is an important aspect of quality of life. There is a link between heart disease and sexual dysfunction. Heart disease lowers the activity or the ability to perform the sexual activity. Sexual problems have a negative impact on quality of life and well-being, and sexual dysfunction is associated with anxiety and depression. The causes of sexual dysfunction are physical changes (the disease), mental changes and adverse reactions from medication. Despite the fact, that several international guidelines recommend that health professionals address sexual function in patients with heart disease, this is rarely done in practice. In Denmark there is no consensus or practice on how or where patients with heart disease and sexual dysfunction should be treated. Some patients are treated with phosphodiesterase type 5 inhibitors and a few referred to sexological clinics. Non-pharmacological rehabilitation interventions such as physical exercise, pelvic floor exercise, and sexual therapy have shown potential beneficial effect on sexual function. However, the effects have not been tested sufficiently, have not been tested in combination, and have never been tested in a Danish population.

Objective: The objective of this trial is to investigate the effect of a comprehensive sexual rehabilitation intervention program, consisting of a psycho-educative component and an exercise-training component plus treatment as usual versus treatment as usual in male patients with impaired sexual function and implantable cardioverter defibrillator or ischemic heart disease.

Design: CopenHeartSF is an investigator-initiated randomised clinical trial with blinded outcome assessment, including two university hospitals, with 1:1 central randomisation to sexual rehabilitation plus usual care versus usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* Male patients above 18 years with sexual dysfunction associated with implantable cardioverter defibrillator or with ischemic heart disease verified by coronary angiography, which have a partner, speaks and understands Danish and provides a written informed consent

Exclusion Criteria:

* Patients at intermediate or high risk according to their cardiovascular status according to guidelines, with diseases in the urinary tract, who exercise intense more than 3 hours a week, patients with neurological or orthopedic deficits which prevent training, patients with cognitive deficits which prevents interviews, and patients who are included in ongoing research prohibiting additional research participation are excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) | 16 week

SECONDARY OUTCOMES:
Psychosocial adjustment to illness scale (PAIS-SR)sexual relationship domain | 16 week

CONTACTS AND LOCATIONS:
Overall Officials: Selina Berg, PhD, Principal Investigator — The Heart Centre, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Hjertecentret, Copenhagen University Hospital, Rigshospitalet, Blegdamsvej 9, Copenhagen, OE, Denmark

REFERENCES:
- [Derived] Palm P, Zwisler AO, Svendsen JH, Thygesen LC, Giraldi A, Jensen KG, Lindschou J, Winkel P, Gluud C, Steinke E, Berg SK. Sexual rehabilitation for cardiac patients with erectile dysfunction: a randomised clinical trial. Heart. 2019 May;105(10):775-782. doi: 10.1136/heartjnl-2018-313778. Epub 2018 Oct 31. PMID 30381319
- [Derived] Johansen PP, Zwisler AD, Hastrup-Svendsen J, Frederiksen M, Lindschou J, Winkel P, Gluud C, Giraldi A, Steinke E, Jaarsma T, Berg SK. The CopenHeartSF trial--comprehensive sexual rehabilitation programme for male patients with implantable cardioverter defibrillator or ischaemic heart disease and impaired sexual function: protocol of a randomised clinical trial. BMJ Open. 2013 Nov 25;3(11):e003967. doi: 10.1136/bmjopen-2013-003967. PMID 24282249